CLINICAL TRIAL: NCT07224243
Title: Impact of Intraoperative Oxygenation Practices on Patient Outcomes
Acronym: IntraOp Ox
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Frederic T Billings IV (Other)
Collaborators: Multicenter Perioperative Outcomes Group (Other); University of Michigan (Other); The Association of University Anesthesiologists (Unknown)
Responsible Party: Sponsor-Investigator, Frederic T Billings IV, Professor of Anesthesiology, Vanderbilt University Medical Center
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 241806
Record Dates: First submitted 2025-10-31; First posted 2025-11-04 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Surgeries Undergoing General Anesthesia
Keywords: Intraoperative oxygenation; oxygen; surgery; anesthesia; mechanical ventilation; organ injury; acute kidney injury; myocardial injury; lung injury; stroke; pragmatic; cluster
MeSH Terms: conditions — Acute Kidney Injury; Lung Injury; Stroke

STUDY DESIGN:
Intervention Model Description: Cluster randomized, cluster crossover
Who Masked: Outcomes Assessor
Masking Description: Outcomes are measured through routine clinical care. The primary statistician is masked to treatment assignments during analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Lower FiO2 (Experimental)
  Interventions: Other: Lower FiO2
- Intermediate FiO2 (Experimental)
  Interventions: Other: Intermediate FiO2
- Higher FiO2 (Experimental)
  Interventions: Other: Higher FiO2

INTERVENTIONS:
Other: Lower FiO2 — FiO₂ 0.21-0.40 or lowest FiO₂ to maintain SpO₂ ≥ 94% during maintenance anesthesia
  Arms: Lower FiO2
Other: Intermediate FiO2 — FiO₂ 0.40-0.80 or lowest FiO₂ to maintain SpO₂ ≥ 94% during maintenance anesthesia
  Arms: Intermediate FiO2
Other: Higher FiO2 — FiO₂ > 0.80 to maintain SpO₂ ≥ 94% during maintenance anesthesia
  Arms: Higher FiO2

SUMMARY:
This multicenter, cluster-randomized, cluster-crossover clinical trial evaluates the impact of three intraoperative FiO2 (Fraction of Inspired Oxygen) oxygenation strategies-lower (FiO₂ 0.21-0.40), intermediate (FiO₂ 0.40-0.80), and higher (FiO₂ 0.80-1.00)-on postoperative organ injury and mortality in adult surgical patients. The trial aims to determine the optimal oxygenation strategy to improve perioperative outcomes.

DETAILED DESCRIPTION:
The Intraop Ox trial will enroll adult patients undergoing surgery with tracheal intubation. Participating hospitals will be randomly assigned (as a unit) to administer one of three oxygenation strategies during maintenance anesthesia (lower FiO₂ [0.21-0.40], intermediate FiO₂ [0.40-0.80], or higher [FiO₂ 0.80-1.00] each period (month). The primary outcome is a composite of organ injury (acute kidney injury, myocardial injury, lung injury, stroke) or death within 30 days. Secondary outcome is 30-day mortality. Exploratory outcomes are individual components of the composite primary endpoint, surgical site infection, length of stay, and hypoxemia. The study is conducted under a waiver of informed consent due to minimal incremental risk of participating and impracticability of obtaining consent in this cluster-randomized design.

ELIGIBILITY:
Inclusion Criteria:

* Patient located in a participating operating room
* Planned surgery includes tracheal intubation

Exclusion Criteria:

* Patient is known to be less than 18 years old
* Patient is known to be pregnant
* Patient is known to be a prisoner.
* Patient is American Society of Anesthesiologists (ASA) classification-6 (i.e., organ donor)
* Patient's planned surgical case includes open heart surgery, defined as surgery on the heart or ascending aorta requiring sternotomy or thoracotomy.
* Patient's planned procedure requires prolonged apnea, bronchoscopy, airway surgery, or one-lung ventilation.
* Patient's planned surgical case includes use of extracorporeal membrane oxygenation (ECMO).
* Patient is known to have a history of bleomycin treatment.
* Patient was enrolled in the trial in the prior 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54000 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Composite of organ injury or in-hospital death within 30 days of surgery | 30 days post-surgery
  This composite outcome measures the number of participants experiencing at least one of the following organ injuries or death within the defined study period:
  * Acute Kidney Injury (AKI), defined according to creatinine based Kidney Disease Improving Global Outcomes criteria, specifically a 0.3 mg/dL or greater increase within 48 hours or a 50% or greater increase from baseline within seven days of surgery.
  * Myocardial injury, defined as >99th percentile of normal based on site-specific troponin assay within 72 hours of surgery.
  * Lung injury, defined using international classification of diseases, ninth revision or tenth revision (ICD-9 or ICD-10) diagnosis codes
  * Stroke, defined using international classification of diseases, ninth revision or tenth revision (ICD-9 or ICD-10) diagnosis codes
  * Death within 30 days of surgery

SECONDARY OUTCOMES:
30-day mortality | 30 days post-surgery
  Death from any cause within 30 days of surgery

OTHER OUTCOMES:
Acute kidney injury | 7 days post-surgery
  Incidence of acute kidney injury (AKI), defined according to creatinine based Kidney Disease Improving Global Outcomes criteria, specifically a 0.3 mg/dL or greater increase from baseline within 48 hours or a 50% or greater increase from baseline within seven days of surgery
Myocardial injury | 72 hours post-surgery
  Myocardial injury, defined as >99th percentile of normal plasma troponin based on site-specific troponin assay within 72 hours of surgery.
Lung injury | 30 days post-surgery
  Lung injury, defined using international classification of diseases, ninth revision or tenth revision (ICD-9 or ICD-10) diagnosis codes
Stroke | 30 days post-surgery
  Stroke, defined using international classification of diseases, ninth revision or tenth revision (ICD-9 or ICD-10) diagnosis codes
Surgical site infection | 30 days post-surgery
  Surgical site infection, defined using National Surgical Quality Improvement Program (NSQIP) criteria and reported to NSQIP and also captured using international classification of diseases (ICD) diagnosis data.
Hospital length of stay | Day of hospital discharge
  Total number of calendar days from the date of surgery to the date of discharge following the index procedure.
Hypoxemia | Perioperative
  Incidence and duration of SpO₂ values < 80% (in minutes) during maintenance anesthesia (from anesthesia induction to anesthesia emergence).

CONTACTS AND LOCATIONS:
Overall Officials: Frederic T Billings, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data cannot be removed from the MPOG servers where they are stored and analysed. We will review requests for data analyses that use individual patient data, but it would have to be performed inside these servers - i.e., IPD cannot not be shared with others.